CLINICAL TRIAL: NCT01650155
Title: Safety, Tolerability, Pharmacokinetics and Early Pharmacodynamics of Single Rising Intravenous and Subcutaneous Doses of BI 1005273 in Healthy Male Volunteers (Randomised, Single-blind, Placebo-controlled Within Dose Groups, Clinical Phase I Study)
Brief Title: Single Rising Dose Study With Intravenous Infusion and Subcutaneous Injection of BI 1005273 in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1294.1; 2011-004987-30 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-07-18; First posted 2012-07-26 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (4):
- BI 1005273 i.v. (Experimental): single dose i.v. infusion
  Interventions: Drug: BI 1005273 i.v.
- BI 1005273 i.v. Placebo (Placebo Comparator): single dose i.v. infusion (Placebo)
  Interventions: Drug: BI 105273 i.v. Placebo
- BI 1005273 s.c. (Experimental): single dose s.c. injection
  Interventions: Drug: BI 1005273 s.c.
- BI 1005273 s.c. Placebo (Placebo Comparator): single dose s.c. injection (Placebo)
  Interventions: Drug: BI 1005273 s.c. Placebo

INTERVENTIONS:
Drug: BI 1005273 s.c. — injection
  Arms: BI 1005273 s.c.
Drug: BI 105273 i.v. Placebo — infusion
  Arms: BI 1005273 i.v. Placebo
Drug: BI 1005273 s.c. Placebo — injection
  Arms: BI 1005273 s.c. Placebo
Drug: BI 1005273 i.v. — infusion
  Arms: BI 1005273 i.v.

SUMMARY:
To investigate the safety and tolerability of BI 1005273 in healthy male volunteers following intravenous (i.v.) infusion of single rising doses and subcutaneous (s.c.) injection. Secondary objectives are the exploration of the pharmacokinetics and early pharmacodynamics of BI 1005273.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects

Exclusion criteria:

1. Any deviation from healthy conditions

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
number (% subjects) with drug-related AEs. | day -21 to day 95

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | day 1 to day 90
AUC0-8 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | day 1 to day 90
AUC0-tz (area under the concentration-time curve of the analyte in the plasma over the time interval from 0 to the last measurable time point of the dose) | day 1 to day 90

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1294.1.1 Boehringer Ingelheim Investigational Site, Berlin, Germany